CLINICAL TRIAL: NCT06986356
Title: The Effects of a Commercially Available High Protein Spoonable on Overnight Recovery From Exercise Training in 18-45 Year-old Male and Females
Brief Title: Spoonable - Overnight Recovery
Acronym: BOLT_PartB
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Danone Nutricia Research (Industry)
Responsible Party: Principal Investigator, Glyn Howatson, Professor Glyn Howatson, Northumbria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: BOLT_PartB_7943
Record Dates: First submitted 2024-10-25; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2024-10

CONDITIONS: Recovery; Muscle Function; Muscle Soreness
MeSH Terms: conditions — Myalgia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test Product: Yoghurt (Experimental): High protein commercially available spoonable yoghurt (1 serving = 45 g protein comprising 3 yoghurt pots totalling 480 g) (Danone Nutricia).
  Interventions: Dietary Supplement: Test product: Yoghurt
- Control Product: Placebo (Jelly) (Placebo Comparator): flavoured water-based placebo jelly (1 serving = 0 g protein comprising 3 jelly pots totalling 480 g).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Test product: Yoghurt — High protein spoonable yoghurt
  Arms: Test Product: Yoghurt
Dietary Supplement: Placebo — Placebo Jelly
  Arms: Control Product: Placebo (Jelly)

SUMMARY:
The key research objective is to examine the effects of a high protein spoonable yoghurt on overnight recovery of muscle function, 12 hours following an exercise session in 18-45-year-old males and females, compared to a control group receiving flavoured waterbased placebo jelly. An additional aim of the study is to explore the effects of the test product vs placebo on muscle function, readiness to exercise and performance in a repeat bout of exercise training at 24 hours following initial exercise training.

DETAILED DESCRIPTION:
This study is a single-blind, randomised, parallel group design. It involves six visits to the laboratory in total; Visit 1) pre-screening and consent; visit 2) questionnaires, anthropometrics, and familiarisation; Visit 3) baseline measures; Visit 4) exercise intervention (exercise session 1); Visit 5) post-exercise morning measures, and Visit 6) exercise intervention (exercise session 2). Participants will be randomised into one of two groups that will receive the following;

1. Test product: High protein spoonable yoghurt (1 serving = 45 g protein comprising 3 yoghurt pots totalling 480 g) (Danone Nutricia).
2. Control product 2: flavoured water-based placebo jelly (1 serving = 0 g protein comprising 3 jelly pots totalling 480 g).

A follow-up communication via telephone will be conducted within 7 days of completion of the final session to ensure there are no adverse effects of participation.

A detailed overview of the research activity that will take place in each session is provided below:

Visit 1: Pre-screening Volunteers will receive information on the study, and they will be familiarised with the requirements for participation and provide written informed consent. Subjects will be requested to complete 3-day food and exercise diaries, comprising of 1 weekend day, 1 rest day, and 1 exercise day within a week of the trial. This will be handed in on Visit 2. Subjects' body height, body mass, body composition, and BMI will be measured.

Visit 2: Familiarisation with the dependent measures and exercise training Volunteers will refrain from physical activity and alcohol consumption 24 hours before each visit and caffeine 12 hours before each visit. Study staff will review physical activity and food diary questionnaires and if eligibility criteria are met, volunteers will continue the trial. Measure of volunteers' body mass, stature and body composition will then be recorded. Next, volunteers will be familiarised with the dependent measures and exercise training session that will be conducted.

Visit 3: Baseline Measures Volunteers will report to the laboratory in the PM in a fed (2-3 hours post prandial) and hydrated state, where baseline measurements of all dependent variables will be taken. Which will include muscle soreness via a visual analogue scale, muscle pain pressure threshold via algometry. Measures of muscle function including Counter Movement Jump (CMJ), Reactive Strength Index (RSI) and Isometric Maximal Voluntary Contraction (iMVC). A venous blood sample will be taken to measure creatine kinase and high sensitivity C-reactive protein.

Following this, volunteers will receive standardised meals for the day of the exercise trial. Standardised meals will provide:

* Total energy (kcals) = BMR (derived via Harris-Benedict) x 1.5 (PAL). Assuming participants will be largely sedentary apart from the exercise session.
* Protein 1g/kg body weight for both groups.
* Carbohydrate - Provide 50% of total energy
* Fat - Remainder of total energy.

Participants will keep their habitual physical activity pattern between visits but not exceeding 4 exercise sessions per week (pro-rata), of which not more than 2 sessions of light resistance exercise sessions can be completed. Any exercise outside of the study will be recorded. Volunteers will be asked to refrain from any strenuous exercise 24 h prior to the first visit and for the duration of the subsequent trial visits (except for that required during the study). Volunteers will record any deviations from the standardised meal plan in a food compliance diary throughout.

Visit 4: First exercise training session Volunteers should consume breakfast before ~8 AM, lunch ~12 PM, and dinner at ~4 PM. Volunteers will attend the study site in the evening, scheduled at least 2 hours after dinner. Study staff will receive completed food compliance diary from volunteers. Volunteers will be asked to complete all dependent measures. This will be followed by the exercise training consisting of an initial warm up, a repeated sprint cycling challenge followed by an exercise circuit that will consist of intermittent high intensity exercises (detailed below) for a period likely to extend approximately 40 minutes. The session will be similar to a high intensity exercise class and the number of repetitions will be recorded in each time window to compare between Visit 4 and 6. Volunteers will wear a heart rate monitor throughout to measure peak and mean heart rate. Immediately after, measures of the participant's lactate concentration and their perceived exertion for the session followed by a further lactate sample at 15 mins. Volunteers will then complete all dependent variables and consume the test product or control product.

The exercise protocol is detailed below and will be repeated in visit 6. Warm up

* Static exercise bike 5 minutes at 1.5 W per Kg Body mass
* Standardised dynamic warm up (~5 minutes of walking lunges, squats & mobility) Cycle Ergometer Repeated Sprint
* 10 x 6s Lode Bike sprints with 30 s (active) recovery Circuit Training 5 rounds with a 30s 1:1 work rest ratio.
* Kettlebell Thrusters (bilateral)
* Squat Jumps (set height from plyometric box)
* Kettlebell Walking Lunge (bilateral) • Kettlebell Swing (single)
* Kettlebell bent-over row
* Sled push 40 m
* Sled pull 40 m
* Farmers walks (bilateral kettlebell) Total time ~60 minutes Notes
* Kettlebell weight to be selected at familiarisation and used throughout (likely ~10-20% BM)
* Sled Row/pull will be a % of BW (TBC - likely 50% BM)

Visit 5: 12-hour overnight recovery following exercise training session 1 The participant will have a standardised breakfast at home ~7 AM and attend the laboratory ~ 2 h after. Participants will attend the study site at ~9 AM. Study staff will receive completed food compliance and study product intake diaries following exercise training 1 session (visit 4). Participants will be asked to complete a Recovery Questionnaire and the Sleep Quality Questionnaire. Participants will complete muscle soreness and pain measures. Study staff will measure volunteers' body mass and draw a blood sample. Next, volunteers will complete all dependent variables. Volunteers will consume a final serving of the study or placebo product in the laboratory when all measures are completed. After the visit volunteers will consume the provided lunch and dinner at home, at ~12PM and ~4PM, respectively.

Visit 6: 24-hour return to training readiness and performance following exercise training session 1 Physiological and performance measures pre- and post-exercise training session 2). Participants will attend the laboratory at least 2 hours after dinner (~18:00). Study staff will receive completed food compliance diary from volunteers between visit 4 and visit 6. Volunteers will be asked to complete the Recovery, Readiness to Exercise, and muscle soreness questionnaires. Study staff will measure volunteers' body mass and draw a blood sample. Then, volunteers will complete all dependent variables. After 10-15 minutes rest, volunteers will complete a second exercise training session, which will be identical to visit 4), wearing a heart rate monitor. Immediately after exercise training session 2, blood lactate concentration will be measured, followed by a further sample at 15 minutes and rate their perceived exertion. Lastly, after these measures volunteers will repeat dependent measures of muscle soreness/pain and muscle function.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 45 years
* Body Mass Index (BMI) ≥ 18.5 and ≤ 29.9 kg/m2
* Written informed consent
* Willingness and ability to comply with the protocol in the opinion of the Investigator
* Judged by the Investigator to be in good health as assessed by a health screening questionnaire
* Currently identifies as the same biological sex as at birth

Exclusion Criteria:

* Any known ongoing medical condition that interferes significantly with absorption and digestion and/or gastrointestinal (GI) function (e.g. inflammatory bowel disease, gastroesophageal reflux disease, celiac disease, diaphragmatic hernia or diaphragmatic surgery, gastric ulcer, gastritis, gall bladder problems, pancreatitis, GI cancer, oesophageal and/or gastric surgery), in opinion of the investigator.
* Known musculoskeletal or soft tissue injury
* Known cardiovascular disease, disease related to the immune system and/or the respiratory system
* Known renal or hepatic failure or known thyroid dysfunction
* Known Diabetes Mellitus type I or type II, insulin resistance or metabolic syndrome
* Any ongoing cancer (except for basal cell carcinoma) and/ or cancer treatment
* Known anaemia or low haemoglobin or low iron status
* Any known bleeding disorder or reaction to withdrawal of blood samples
* Use of oral and systemic use of prokinetics, laxatives, antidiarrheals, anticoagulants within 2 weeks prior to screening
* Use of systemic antibiotics within 4 weeks prior to screening
* Any known allergies or intolerances to ingredients of the study product, i.e. cow's milk allergies, lactose intolerance
* Adherence to a strict dietary regime (e.g. vegetarian/ vegan/ paleo/ketogenic/intermittent fasting/ high protein diet (>1.6 g/kg body weight/day) or a weight loss program)
* Use of any nutritional supplements or additional protein supplements or nutritional support within 4 weeks prior to screening
* Falling below or exceeding the classification of Tier 1 or Tier 2 (McKay et al 2022, IJSPP. 17, 317-331). Ranging from minimum of meeting WHO guidelines for physical activity up to training ~3 times per week and local level representation in a sport.
* Known pregnancy and/or lactation
* Current smoking or stopped smoking for <1 month prior to screening (except for incidental smoking of ≤3 cigarettes/cigars/pipes per week on average in the last month)
* Average alcohol use of >21 glasses* per week for men or >14 glasses per week for women (on average during the last 6 months) or drug/ medicine abuse in opinion of the investigator
* Participation in any other clinical study with investigational or marketed products concomitantly or within 4 weeks before screening.
* Major medical or surgical event requiring hospitalization within the preceding 3 months and/or scheduled in the period of study participation relevant in the opinion of the Investigator

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2025-06-13 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Muscle Function (Maximal voluntary contraction) | Testing will occur over a two week period (from visit 2-6).This measure will be taken at baseline (visit 3), before and after exercise session 1 (visit 4), 12 hours after exercise session 1 (visit 5) and before and after exercise session 2 (visit 6).
  The change from baseline in muscle function (measured via quadriceps maximum voluntary contraction; MVC) 12 hours after exercise session 1. This measurement reflect the ability for the intervention group to recovery faster or have less decrements in function. MVC will be assessed with a bespoke dynamometer (three efforts will be performed).
Muscle Function (Jump Height) | Testing will occur over a two week period (from visit 2-6). This measure will be taken at baseline (visit 3), before and after exercise session 1 (visit 4), 12 hours after exercise session 1 (visit 5) and before and after exercise session 2 (visit 6).
  The change from baseline in muscle function (assessed by vertical jump height) 12 h after exercise session 1. This measurement reflect the ability for the intervention group to recovery faster or have less decrements in function. Vertical jump height will be assessed by a countermovement jump (CMJ).
Muscle Function (Reactive Strength Index) | Testing will occur over a two week period (from visit 2-6). This measure will be taken at baseline (visit 3), before and after exercise session 1 (visit 4), 12 hours after exercise session 1 (visit 5) and before and after exercise session 2 (visit 6).
  The change from baseline in muscle function (assessed by reactive strength index; RSI) 12 h after exercise session 1. This measurement reflect the ability for the intervention group to recovery faster or have less decrements in function. RSI will be assessed by three drop jumps (average height and ground contact time [cm/m, %change]).

SECONDARY OUTCOMES:
Muscle Function (MVC 24 h post) | Testing will occur over a two week period (from visit 2-6).This measure will be taken at baseline (visit 3), before and after exercise session 1 (visit 4), 12 hours after exercise session 1 (visit 5) and before and after exercise session 2 (visit 6).
  The change from baseline in muscle function (measured via quadriceps maximum voluntary contraction; MVC) 24 h after exercise session 1. This measurement reflect the ability for the intervention group to recovery faster or have less decrements in function. MVC will be assessed with a bespoke dynamometer (three efforts will be performed).
Muscle Function (Jump Height 24 h post) | Testing will occur over a two week period (from visit 2-6).This measure will be taken at baseline (visit 3), before and after exercise session 1 (visit 4), 12 hours after exercise session 1 (visit 5) and before and after exercise session 2 (visit 6).
  The change from baseline in muscle function (assessed by vertical jump height) 24 h after exercise session 1. This measurement reflect the ability for the intervention group to recovery faster or have less decrements in function. Vertical jump height will be assessed by a countermovement jump (CMJ).
Muscle Function (RSI 24 h post) | Testing will occur over a two week period (from visit 2-6). This measure will be taken at baseline (visit 3), before and after exercise session 1 (visit 4), 12 hours after exercise session 1 (visit 5) and before and after exercise session 2 (visit 6).
  The change from baseline in muscle function (assessed by reactive strength index; RSI) 24 h after exercise session 1. This measurement reflect the ability for the intervention group to recovery faster or have less decrements in function. RSI will be assessed by three drop jumps (average height and ground contact time [cm/m, %change]).
Perceived Recovery | Testing will occur over a two week period (from visit 2-6). This measure will be taken at baseline (visit 3), before exercise session 1 (visit 4), 12 hours after exercise session 1 (visit 5) and before exercise session 2 (visit 6).
  The change from baseline in perceived recovery [score] assessed by a recovery questionnaire across the experimental period post-exercise training session 1, between groups
Subjective Muscle Soreness | Testing will occur over a two week period (from visit 2-6). This measure will be taken at baseline (visit 3), before and after exercise session 1 (visit 4), 12 hours after exercise session 1 (visit 5) and before and after exercise session 2 (visit 6).
  The change in subjective pain as assessed by a visual analogue scale (0 - 200mm scale, with extremes either end, 0 referring to no pain at all, 200 referring to extreme pain) over time between groups.
Muscle Pain Pressure | Testing will occur over a two week period (from visit 2-6). This measure will be taken at baseline (visit 3), before and after exercise session 1 (visit 4), 12 hours after exercise session 1 (visit 5) and before and after exercise session 2 (visit 6).
  The change in pain pressure threshold using algometry of the quadriceps, from baseline and during the time course of the study.
Sprint Performance (PPO) | Testing for this measure will occur 48 hour period (two consecutive evening exercise sessions). This measure will be assessed during exercise session 1 (visit 4) and session 2 (visit 6).
  The change in repeated sprint cycle performance (peak power output; PPO, measured by watts), between the two groups.
Sprint Performance (av. PO) | Testing for this measure will occur 48 hour period (two consecutive evening exercise sessions). This measure will be assessed during exercise session 1 (visit 4) and session 2 (visit 6).
  The change in repeated sprint cycle performance (mean; average, power output, measured by watts), between the two groups
Sprint Performance (fatigue index) | Testing for this measure will occur 48 hour period (two consecutive evening exercise sessions). This measure will be assessed during exercise session 1 (visit 4) and session 2 (visit 6).
  The change in repeated sprint cycle performance (fatigue index, quantified by percentage decrease between repetitions of sprints), between the two groups
Readiness to Train | Testing will occur over a two week period (from visit 2-6). This measure will be taken at baseline (visit 3), before and after exercise session 1 (visit 4), 12 hours after exercise session 1 (visit 5) and before and after exercise session 2 (visit 6).
  The change from baseline in perceived readiness to train assessed by the Return to Readiness Questionnaire [visual analogue scale] at 24 hours post-exercise training session 1, between the groups. The scale is 0-100mm, where 0 refers to 'not at all ready to train' and 100 refers to 'extremely ready to train'.
Marker of muscle damage (CK) | Testing will occur over a two week period (from visit 2-6). This measure will be taken at baseline (visit 3), before exercise session 1 (visit 4), 12 hours after exercise session 1 (visit 5) and before exercise session 2 (visit 6).
  The change from baseline over time between groups for muscle damage (serum creatine kinase (CK) [IU/L]).
Marker of inflammation (hs-CRP) | Testing will occur over a two week period (from visit 2-6). This measure will be taken at baseline (visit 3), before exercise session 1 (visit 4), 12 hours after exercise session 1 (visit 5) and before exercise session 2 (visit 6).
  The change from baseline over time between groups for inflammation (serum C-reactive protein (hsCRP) [mg/L]).
Other performance parameters (peak HR) | Testing for this measure will occur 48 hour period (two consecutive evening exercise sessions). This measure will be assessed during exercise session 1 (visit 4) and session 2 (visit 6).
  The changes in performance parameters during exercise sessions 1 and 2, variables include peak heart rate [BPM] during exercise training session 1 and 2.
Other performance parameters (mean HR) | Testing for this measure will occur 48 hour period (two consecutive evening exercise sessions). This measure will be assessed during exercise session 1 (visit 4) and session 2 (visit 6).
  The changes in performance parameters during exercise sessions 1 and 2, variables include mean heart rate [BPM] during exercise training session 1 and 2.
Other performance parameters (RPE) | Testing for this measure will occur 48 hour period (two consecutive evening exercise sessions). This measure will be assessed during exercise session 1 (visit 4) and session 2 (visit 6).
  The changes in other performance parameters during exercise sessions 1 and 2 such as exercise session rating of perceived exertion (RPE). The scale used will be the Borg (6-20) RPE scale, where 6 refers to 'no exertion' and 20 refers to 'maximal exertion'.
Other performance parameters (lactate) | Testing for this measure will occur 48 hour period (two consecutive evening exercise sessions). This measure will be assessed during exercise session 1 (visit 4) and session 2 (visit 6).
  The changes in other performance parameters during exercise sessions 1 and 2, such as pre and post-exercise lactate (immediately post and 15 mins-post).
Perceived Sleep Questionnaire | Testing will occur over a two week period (from visit 2-6). This measure will be taken at baseline (visit 3), before exercise session 1 (visit 4) and 12 hours after exercise session 1 (visit 5).
  The change from baseline in perceived sleep [score] assessed by a sleep questionnaire across the experimental period post-exercise training session 1, between groups. The score is 1-5, where 1 refers to a 'very poor' quality of sleep and 5 refers to 'very good' quality of sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Glyn Howatson, Principal Investigator — Northumbria University
Locations (1):
- Northumbria University, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: No